CLINICAL TRIAL: NCT07196137
Title: Comparing the Effect of Laryngeal Tube Suction (LTS) and Air-Q sp3G Laryngeal Mask Airway (LMA) Use on Gastric Insufflation and Volume Using Ultrasound
Brief Title: Comparing the Effect of LTS and Air-Q sp3G LMA Use on Gastric Insufflation Using Ultrasound
Status: Completed | Type: Observational
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Sponsor
Other Study IDs: E2-25-11500
Record Dates: First submitted 2025-08-19; First posted 2025-09-29 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2025-09

CONDITIONS: Laryngeal Masks Comparison; Elective Surgeries; Gastric Ultrasonography; Gastric Insufflation
Keywords: Laryngeal Mask; Airway Management; Ultrasonography; Child

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- AIRQ: After obtaining consent, patients will be asked to choose their airway device using a sealed envelope method. The patients' demographic data and ASA scores will be recorded. Gastric antrum diameters will be recorded at the beginning of the case, before induction. After the airway device is placed, the antrum diameters will be recorded. The antrum diameters will be recorded again after the surgery is complete, before the airway device is removed. Mechanical ventilator settings will be recorded. To ensure standardization, the tidal volume will be set to 7 ml per kg. No PEEP will be applied. Volume-controlled ventilation will be used. The lowest intraoperative saturation and the highest peak pressure that occurred will be recorded.The cuff pressure will be recorded after being inflated with the recommended volume. The time taken for airway device placement (the time from when it is picked up until Endtidal CO2 is observed) and any failed placements will be recorded.
- LTS: After obtaining consent, patients will be asked to choose their airway device using a sealed envelope method. The patients' demographic data and ASA scores will be recorded.
  Gastric antrum diameters will be recorded at the beginning of the case, before induction. After the airway device is placed, the antrum diameters will be recorded. The antrum diameters will be recorded again after the surgery is complete, before the airway device is removed.
  Mechanical ventilator settings will be recorded. To ensure standardization, the tidal volume will be set to 7 ml per kg. No PEEP will be applied. Volume-controlled ventilation will be used. The lowest intraoperative saturation and the highest peak pressure that occurred will be recorded.The cuff pressure will be recorded after being inflated with the recommended volume.
  The time taken for airway device placement (the time from when it is picked up until Endtidal CO2 is observed) and any failed placements will be recorded.

SUMMARY:
The primary objective of the study is to evaluate gastric insufflation during the use of two different airway devices (Laringeal Tube Suction and Air Q sp3G Laryngeal Mask.

The secondary objectives of the study are to assess these two airway devices in terms of perioperative complications.

DETAILED DESCRIPTION:
During general anesthesia, various devices are used to secure the airway. Supraglottic airway devices (SGAs) are among these and are used safely for short surgical procedures. Although SGAs are used to provide an easy and safe airway, none of them seal the trachea and ventilate only the lungs in the way that endotracheal intubation (ETT) does. Positive pressure ventilation provided at the supraglottic level cannot prevent air from escaping into the esophagus and, consequently, the stomach. Gastric distension is associated with perioperative complications such as nausea, vomiting, and aspiration, and is considered an undesirable condition by anesthesiologists.

The study aims to compare the Laryngeal Tube Suction and the Air Q sp3G Laryngeal Mask in terms of gastric insufflation. By measuring the diameters of the gastric antrum and recording their changes throughout the case, this study intend to evaluate the effectiveness and reliability of the two airway devices.

ASA (American Society of Anesthesiologist) I-III class pediatric patients between the ages of 1-12 who will undergo elective surgery under general anesthesia will be included in the study. Randomisation will be done with a sealed envelope. The blinded researcher will collect and record data without knowing which airway device was chosen. Blind researcher will do gastric ultrasound measurements with Butterfly IQ+ ultrasound. Another researcher will insert the airway device and after insertion patients head will be covered, this researcher will not involve during data collection. After the data is collected, the airway device releated data will be recorded by non-blind researcher seperately.

ELIGIBILITY:
Inclusion criteria:

Patients with an ASA score of I-III for whom a supraglottic airway (SGA) is planned.

Operation time less than 2 hours. Patients who have read and accepted the informed consent form. Patients between the ages of 1 and 12, or their guardians, will be included in the study.

Exclusion criteria:

Patients who do not meet perioperative fasting criteria. Patients whose stomachs are not considered empty during the initial gastric ultrasound.

Patients with a known difficult airway. Patients with oropharyngeal or laryngeal anomalies. Patients who require the use of neuromuscular blockers. Patients with a history of a previously failed SGA placement. Patients with known reflux. Patients who do not give consent will not be included in the study.

Ages: 1 Year to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: ASA I-III class, ages between 1-12, patients who will undergo elective surgery under standard general anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 101 (Actual)
Dates: Start 2025-09-29 (Actual); Primary Completion 2026-01-02 (Actual); Study Completion 2026-01-29 (Actual)

PRIMARY OUTCOMES:
Gastric Antral Cross Sectional Area (T0) | Just before anesthesia induction
  First gastric measurement: Before anesthesia induction gastric ultrasound will be done and gastric antrum cross sectional area will be recorded by blinded researcher
Gastric Antral Cross Sectional Area (T1) | Right after the SGA is placed following anesthesia induction.
  Second gastric measurement: after anesthesia induction and before the start of surgery gastric ultrasound will be done and gastric antrum cross sectional area will be recorded by blinded researcher
Gastric Antral Cross Sectional Area (T2) | Just before the end of anesthesia, after the surgery is completed
  Third measurement: Just before the end of anesthesia, after the surgery is completed gastric ultrasound will be done and gastric antrum cross sectional area will be recorded by blinded researcher.

SECONDARY OUTCOMES:
LTS Cuff Pressure Measurement | Just after inserting a Laryngeal Tube Suction
  If the choosen airway device is an LTS, after inserting LTS a cuff pressure measurement will be done by nonblind researcher. For masking the device that used even if a measurement is not taken, it will be treated as if it were.
Maximum Airway Pressure (PPeak) | Intraoperative
  The highest pressure measured by the mechanical ventilator will be recorded.
Minimum Saturation | Intraoperative
  The lowest measured saturation value.
Spasm | Intraoperative and/or postoperative 2 hours
  Incidence of spasm
The time taken for airway device placement and failed placement | Intraoperative
  The time from the moment the airway device is touched until end-tidal CO2 is detected (Second)
Postoperative Sore Throat | Postoperative 2 hours
  Incidence of sore throat assessed by direct questioning
Postoperative Nausea and Vomitting | Postoperative 2 hours
  Incidence of post operative nausea and vomitting assessed by direct questioning
Presence of blood on the supraglottic airway | Just after removing the SGA
  Nonblinded researcher will check if there is blood contamination on the SGA after removing it.
Postoperative Cough | Postoperative 2 hours
  Incidence of Cough assessed by direct questioning or physical examination
Need for nebulized medications or cool mist. | Postoperative 2 hours
  Need for nebulized medications or cool mist for spasm or cough

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Bilkent City Hospital Department of Anesthesiology and Reanimation, Ankara, Çankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chandrakar S, Sreevastava DK, Bhasin S, Dhar M. Comparison of laryngeal tube suction II and proseal LMA in pediatric patients, undergoing elective surgery. Saudi J Anaesth. 2017 Oct-Dec;11(4):432-436. doi: 10.4103/sja.SJA_418_17. PMID 29033724
- [Background] Gasteiger L, Ofner S, Stogermuller B, Ziegler B, Brimacombe J, Keller C. Randomized crossover study assessing oropharyngeal leak pressure and fiber optic positioning : Laryngeal Mask Airway Supreme versus Laryngeal Tube LTS II size 2 in non-paralyzed anesthetized children. Anaesthesist. 2016 Aug;65(8):585-9. doi: 10.1007/s00101-016-0192-1. PMID 27380049
- [Background] Genzwuerker HV, Finteis T, Slabschi D, Groeschel J, Ellinger K. Assessment of the use of the laryngeal tube for cardiopulmonary resuscitation in a manikin. Resuscitation. 2001 Dec;51(3):291-6. doi: 10.1016/s0300-9572(01)00410-5. PMID 11738781
- [Background] Scheller B, Schalk R, Byhahn C, Peter N, L'Allemand N, Kessler P, Meininger D. Laryngeal tube suction II for difficult airway management in neonates and small infants. Resuscitation. 2009 Jul;80(7):805-10. doi: 10.1016/j.resuscitation.2009.03.029. Epub 2009 May 2. PMID 19410354
- [Background] Katzenschlager S, Mohr S, Kaltschmidt N, Peterstorfer F, Weilbacher F, Gunther P, Ries M, Weigand MA, Popp E. Laryngeal mask vs. laryngeal tube trial in paediatric patients (LaMaTuPe): a single-blinded, open-label, randomised-controlled trial. Eur J Emerg Med. 2025 Apr 1;32(2):123-130. doi: 10.1097/MEJ.0000000000001178. Epub 2024 Sep 12. PMID 39264430